CLINICAL TRIAL: NCT04678375
Title: Classification of Retinal Diseases by Artificial Intelligence
Brief Title: Artificial Intelligence for Detecting Retinal Diseases
Status: Completed | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Beijing Tulip Partner Technology Co., Ltd, China (Unknown)
Responsible Party: Sponsor
Other Study IDs: AI in retinal diseases
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2018-06

CONDITIONS: Artificial Intelligence; Retinal Diseases
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retinal diseases diagnosed by artificial intelligence algorithm: Retinal diseases diagnosed by artificial intelligence algorithm
  Interventions: Diagnostic Test: Retinal diseases diagnosed by artificial intelligence algorithm

INTERVENTIONS:
Diagnostic Test: Retinal diseases diagnosed by artificial intelligence algorithm — An artificial intelligence algorithm was applied to diagnose referral diabetes retinopathy, referral age-related macular degeneration, referral possible glaucoma, pathological myopia, retinal vein occlusion, macular hole, macular epiretinal membrane, hypertensive retinopathy, myelinated fibers, retinitis pigmentosa and other retinal lesions from fundus photography.

SUMMARY:
The objective of this study is to apply an artificial intelligence algorithm to diagnose multi retinal diseases from fundus photography. The effectiveness and accuracy of this algorithm was evaluated by sensitivity, specificity, positive predictive value, negative predictive value, and area under curve.

DETAILED DESCRIPTION:
The objective of this study is to apply an artificial intelligence algorithm to diagnose referral diabetes retinopathy, referral age-related macular degeneration, referral possible glaucoma, pathological myopia, retinal vein occlusion, macular hole, macular epiretinal membrane, hypertensive retinopathy, myelinated fibers, retinitis pigmentosa and other retinal lesions from fundus photography. The effectiveness and accuracy of this algorithm was evaluated by sensitivity, specificity, positive predictive value, negative predictive value, area under curve, and F1 score.

ELIGIBILITY:
Inclusion Criteria:

* fundus photography around 45° field which covers optic disc and macula
* complete identification information

Exclusion Criteria:

* insufficient information for diagnosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is derived from an anonymous database that contains health examination results of the general population.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Area under curve | 1 week
  We used the receiver operating characteristic (ROC) curve and area under curve to examine the ability of this artificial intelligence algorism recognition and classification of retinal diseases.
Sensitivity and specificity | 1 week
  We used sensitivity and specificity to examine the ability of this artificial intelligence algorism recognition and classification of retinal diseases.
Positive predictive value, negative predictive value | 1 week
  We used positive predictive value and negative predictive value to examine the ability of this artificial intelligence algorism recognition and classification of retinal diseases.
F1 score | 1 week
  We used F1 score to examine the ability of this artificial intelligence algorism recognition and classification of retinal diseases.

SECONDARY OUTCOMES:
Systemic biomarkers and diseases | 1 week
  Using medical records as the gold standard, we test the accuracy of this artificial intelligence algorism recognition and classification of systemic biomarkers and diseases: age, sex, blood pressure, blood hemoglobin, cardiovascular diseases, thyroid function and kidney function.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Wei, Study Chair — Beijing Tongren Hospital
Locations (1):
- Wen-Bin Wei, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No